CLINICAL TRIAL: NCT03741075
Title: Topical Tranexamic Acid Plus Bilateral Uterine Artery Ligation During Hemorrhagic Cesarean Delivery for Complete Placenta Previa: a Randomized Double-blind Controlled Trial
Brief Title: Topical Tranexamic Acid Plus Bilateral Uterine Artery Ligation During Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/198/18
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cesarean Section Complications
Keywords: placenta previa; tranexamic acid; uterine artery ligation
MeSH Terms: conditions — Placenta Previa | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: The current study was a double-blind randomized controlled trial will be conducted at a tertiary University Hospital
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which was used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUAL plus placebo (Active Comparator): bilateral uterine artery ligation (BUAL) after delivery of the fetus which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures plus 200 ml saline topical application to placental bed
  Interventions: Procedure: BUA; Drug: placebo
- BUAL plus topical tranexamic acid (Experimental): bilateral uterine artery ligation (BUAL) after delivery of the fetus which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures plus topical application of 20ml saline contains 2 gm tranexamic acid
  Interventions: Procedure: BUA; Drug: topical tranexamic acid

INTERVENTIONS:
Procedure: BUA — bilateral uterine artery ligation (BUAL) after delivery of the fetus which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures
  Other Names: Active Comparator
Drug: topical tranexamic acid — topical application of 200ml saline contains 2 gm tranexamic acid to the placental bed after delivery of the fetus which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures
  Other Names: active comparator
  Arms: BUAL plus topical tranexamic acid
Drug: placebo — topical application of 200ml saline to the placental bed after delivery of the fetus which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures
  Other Names: Placebo to tranexamic acid
  Arms: BUAL plus placebo

SUMMARY:
Placenta previa (PP) is an obstetric condition that is closely linked with massive obstetric hemorrhage with a varied incidence about once in every 200 live births. It is considered one of the causes of the increased need for blood transfusion and cesarean hysterectomy. PPH due to PP typically starts during cesarean section (CS) in the placental bed, at the lower uterine segment mostly after placental separation. Proceeding for cesarean hysterectomy can be the only effective line of management in spite of the associated high morbidity rate.

Various conservative measures have been developed to avoid hysterectomy and preserve fertility in patients with PP. Bilateral Uterine artery ligation (BUAL) is one of the reported surgical procedures carried out in these cases as it is easy and quick. It can be used alone or with adjunctive measures with a fair success rate. The aim is to reduce the blood supply to the uterus and to prevent postpartum hemorrhage.

Tranexamic acid is a lysine analog which acts as an antifibrinolytic via competitive inhibition of the binding of plasmin and plasminogen to fibrin. The rationale for its use in the reduction of blood loss depending on the implication of the coagulation and fibrinolysis processes implicated in the control of PPH. However, concerns about possible thromboembolic events with parenteral administration of TA have stimulated increasing interest in its topical use.

DETAILED DESCRIPTION:
Study inclusion criteria will be women undergoing elective cesarean delivery for complete placenta previa which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures Eligible participants were allocated to one of two groups. Group (I): patients managed by bilateral uterine artery ligation (BUAL) after delivery of the fetus which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures. Group (II): patients received 1 gm TA (2 ampoules of Capron® 500 mg /5 ml; Cairo, Egypt) topically applied to the placental bed plus BUA when not respond to uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing elective cesarean delivery for complete placenta previa which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures

Exclusion Criteria:

* patients with the high possibility of morbid adherent placenta
* those presented with severe antepartum hemorrhage
* Patients with cardiac, hepatic, renal, or thromboembolic disease;
* hypersensitivity or contraindications of use of tranexamic acid
* patient refuses to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women undergoing elective cesarean delivery for complete placenta previa which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with postpartum hemorrhage | 6 hours post operative
  number pf participants with blood loss > 1000ml

SECONDARY OUTCOMES:
intraoperative blood loss | during the operation
  amount of blood loss during cesarean section
The number of participant needed for blood transfusion | 24 hours post operative
  Calculation of the number of participant needed for blood transfusion
The number of participant needed of extra surgical maneuvers | 24 hours post operative
  Calculation of the number of participant needed of extra surgical maneuvers like internal iliac artery ligation

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided